CLINICAL TRIAL: NCT01971736
Title: Randomized-controlled Split-face Treatment of Facial Rhytids and Laxity in Asians Using Long-pulse 1064nm Laser
Brief Title: Efficacy of Long Pulsed 1064nm Laser for Facial Skin Tightening
Status: Completed | Type: Observational
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R079h/55
Record Dates: First submitted 2013-03-07; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Skin Tightening; Skin Laxity; Wrinkle Reduction
Keywords: 1064nm YAG laser; laxity; rhytides; asian
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1064nm laser, laxity: split-face single-blind randomized placebo-controlled trial evaluating improvement in facial skin laxity of the side of the face with placebo versus laser

SUMMARY:
We study the efficacy of 1 pass of stacking pulses of long pulse 1064nm laser on the face for skin tightening immediately post laser and 3 months follow up.

DETAILED DESCRIPTION:
To study the efficacy on facial skin tightening and wrinkle reduction after a single pass of double stacking pulses of long pulse 1064nm laser on the face in skin types III-V immediately post procedure and at 3 months. The study is a split-face placebo-controlled single-blind study.

ELIGIBILITY:
Inclusion Criteria:

* ages 35-60 years

Exclusion Criteria:

1. History of skin malignancy
2. Patients on immunosuppression
3. Patients with other known internal malignancy
4. Patients with malnutrition, vitamin or mineral insufficiency
5. Patients on colchicine, penicillamine
6. Patients with weight loss 7.5% of usual body weight within 3 months
7. history of botulinum toxin injection within 6 months
8. history of facial filler injection within 1year

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy adults with visble signs of aging
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pinyapat - Kanechorn-Na-Ayuthaya, M.D., Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Dept. of dermatology, Phramongkutklao hospital, Bangkok, Thailand